CLINICAL TRIAL: NCT04216654
Title: The Role of Helicobacter Pylori in Microalbuminuria in Type 2 Diabetic Patients
Brief Title: Role of Helicobacter Pylori in Microalbuminuria
Status: Completed | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Hosam Mohammad Ahmad, Dr., Minia University
Other Study IDs: H.pylori and microalbuminuria
Record Dates: First submitted 2019-12-31; First posted 2020-01-03 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Microalbuminuria Due to Type 2 Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group(A): 52 cases of type 2 diabetic patients.They have +ve Serum antibody and Stool antigen specific for Helicobacter pylori.
  Interventions: Diagnostic Test: ELISA (enzyme-linked immunosorbent assay)
- Group(B): 36 cases of type 2 diabetic patients. They have +ve Serum antibody and -ve Stool antigen-specific for Helicobacter pylori.
  Interventions: Diagnostic Test: ELISA (enzyme-linked immunosorbent assay)
- Group(C): 112 cases of type 2 diabetic patients. They have -ve Serum antibody and Stool antigen-specific for Helicobacter pylori.
  Interventions: Diagnostic Test: ELISA (enzyme-linked immunosorbent assay)

INTERVENTIONS:
Diagnostic Test: ELISA (enzyme-linked immunosorbent assay) — ELISA Principle. Enzyme-linked Immunosorbent Assays (ELISAs) combine the specificity of antibodies with the sensitivity of simple enzyme assays, by using antibodies or antigens coupled to an easily-assayed enzyme. ELISAs can provide a useful measurement of antigen or antibody concentration.

SUMMARY:
The aim of this study is to:

1. Investigate a possible association between microalbuminuria and infection by H. pylori in type 2 diabetic patients.
2. Investigate the effect of previous and active infection of H. pylori on microalbuminuria in type 2 diabetic patients.

DETAILED DESCRIPTION:
Helicobacter pylori, previously known as Campylobacter pylori, is a gram-negative, microaerophilic bacterium usually found in the stomach. It was identified in 1982 by Australian scientists Barry Marshall and Robin Warren, who found that it was present in a person with chronic gastritis, gastric ulcers and conditions not previously believed to have a microbial cause. It is also linked to the development of duodenal ulcers and stomach cancer. However, over 80% of individuals infected with the bacterium are asymptomatic, and it may play an important role in the natural stomach ecology. [1] More than 50% of the world's population have H. pylori in their upper gastrointestinal tract. [2] Infection is more common in developing countries than Western countries. [3] H. pylori's helical shape (from which the genus name derives) is thought to have evolved to penetrate the mucoid lining of the stomach. [4, 5] Microalbuminuria, which is defined as an increased urinary albumin to creatinine ratio (UACR) of 30-300 μg/mg .[15] Has been known to be a strong predictor of the development of diabetic nephropathy. [16] It has also been demonstrated that microalbuminuria is a risk factor for cardiovascular disease in the general and diabetic populations. [17-19] and the increased urinary leakage of albumin reflects vascular damage, i.e., endothelial dysfunction or low grade chronic inﬂammation. [20] In addition, some studies have reported a relationship between microalbuminuria and metabolic syndrome, suggesting that insulin resistance underlies the pathogenesis of microalbuminuria. [21-23]

ELIGIBILITY:
Inclusion Criteria:

* Age >45 years and absence of any sever illness.

Exclusion Criteria:

* 1. Those receiving anti-ulcer treatment in the last three months and still receiving proton-pump inhibitors (PPI) or H2 receptor blockers.

  2. Diabetic patients with poor glucose regulation diagnosed previously and detected in laboratory parameters as having diabetic nephropathy.

  3. Those have diabetic retinopathy, neuropathy. 4. Those have renal impairment or known to have renal disease. 5. Those have any primary kidney disease. 6. Those have any systemic disease that my affect the kidney. 7. Those have lupus erythematosus, rheumatoid or other immunological disease. 8. Those have any chronic illness that may affect the kidney 9. Those have urinary tract infections or renal stones. 10. Those may have proteinuria due to any other cause. 11. Heavy exercise, excessive protein ingestion, fluid overload, increase the urinary protein excretion discarded from the study.

  12. Those have chronic liver disease. 13. Those have heart failure. 14. Hypertensive patients. 15. Diabetics having >120 mmHg systolic blood pressure and >85 mmHg diastolic blood pressure.

  16. Those have malignancy. 17. Those with inflammatory disease, those obliged to continue antibiotic treatment for various reasons 18. Smokers 19. Those not providing consent for the study

Ages: 45 Years to 64 Years | Sex: All
Age Groups: Adult
Study Population: 200 adult Type 2 Diabetic patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
association between microalbuminuria and infection by H. pylori in type 2 diabetic patients. | baseline time
  Measure the urinary albumin to creatinine ratio (UACR) to estimate the presence of Microalbuminuria in type 2 diabetic patients among H. pylori-infected, old infected and non infected patients

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo, Cairo, Egypt

REFERENCES:
- See also: book — https://books.google.com.eg/books?hl=ar&lr=&id=UkupDgAAQBAJ&oi=fnd&pg=PT20&dq=Brunette,+G.W.,+CDC+Yellow+Book+2018:+health+information+for+international+travel.+2017:+Oxford+University+Press.&ots=fx0OkjWECM&sig=cP_G5SrjKdNGKESQoJn-lb5WOBc&redir_esc=y#v=onepage&q=Brunette%2C%20G.W.%2C%20CDC%20Yellow%20Book%202018%3A%20health%20information%20for%20international%20travel.%202017%3A%20Oxford%20University%20Press.&f=false
- See also: pdf file — https://pdfs.semanticscholar.org/f58f/54338a7ec5f86920ecb5a900f63669bb7510.pdf